CLINICAL TRIAL: NCT00424450
Title: Assessment of Revascularization Effects in Peripheral Arterial Disease Using Contrast Ultrasound Tissue Perfusion Imaging (REVASC-PI)
Brief Title: Assessment of Bypass Surgery and Balloon Angioplasty Effects in Peripheral Arterial Disease Using Contrast Ultrasound
Status: Completed | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Daniel Duerschmied, Attending, University Hospital Freiburg
Other Study IDs: C01-2006
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Peripheral Arterial Disease
Keywords: contrast ultrasound; muscle perfusion
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PAD patients: 30 PAD patients
  Interventions: Procedure: lower limb artery bypass surgery; Procedure: percutaneous angioplasty (PTA)

INTERVENTIONS:
Procedure: lower limb artery bypass surgery — bypass of severe atherosclerotic vascular lesion
  Other Names: half of the included PAD patients undergo surgery
Procedure: percutaneous angioplasty (PTA) — PTA of severe atherosclerotic lesion
  Other Names: half of included PAD patients undergo PTA

SUMMARY:
Contrast ultrasound perfusion imaging (CUPI) is a novel tool for the assessment of muscle perfusion deficits in peripheral arterial disease (PAD). In this study we want to examine the effect of bypass surgery and balloon angioplasty on the calf muscle blood supply. We hope find a new way of quantifying success or failure of invasive treatment strategies.

DETAILED DESCRIPTION:
Contrast ultrasound perfusion imaging (CUPI) was developed at the University Hospital of Freiburg, Germany in 2005 for the assessment of skeletal muscle perfusion deficits in peripheral arterial disease (PAD). It has been reported previously by the investigators that the contrast agent wash-in is significantly prolonged in PAD with respect to the extent of disease and with respect to the degree of collateralization.

The goal of this study is to examine the effect of revascularization procedures on muscular perfusion in 15 PAD patients undergoing lower limb artery bypass surgery and 15 PAD patients undergoing percutaneous angioplasty (PTA) before and after intervention. Based on the data from a pilot study, a power calculation for an alpha = 5% with a power of 80% and an assumed standard deviation of 10 s yielded a necessary patient number of 29 per group to detect a decrease in wash-in time of 7.5 s. In this intra-individual comparison we aim to compare 30 patients pre with the same 30 patients post revascularization.

We hypothesize 1) that the contrast agent wash-in in the target muscle will significantly improve after revascularization and 2) that standard non-invasive tests such ankle-brachial index (ABI) will not correlate with the CUPI findings. The results of this trial will help to further understand the diagnostic accuracy of CUPI in quantifying limb muscle perfusion deficits.

Patients with symptomatic PAD and an indication for revascularization will undergo CUPI less than 8 weeks prior and less than 3 weeks after the revascularization procedure. A second follow-up CUPI examination is performed 3 - 6 months after the revascularization procedure.

ELIGIBILITY:
Inclusion Criteria:

* male or females > 18 years old
* PAD Fontaine stages IIb, III or IV
* conventional angiography or magnetic resonance angiography
* a severe lesion (≥80% stenosis with a peak velocity ratio intrastenotic / prestenotic ≥4.0 in Duplex ultrasound or occlusion) has to be present in the common or external iliac, common or superficial femoral, popliteal or one or more infrapopliteal arteries, which is accessible to revascularization
* indication for revascularization, i.e. lower limb artery bypass surgery or PTA (based on the treating physician's decision)
* revascularization appointed within the next 6 weeks of study inclusion
* patients, who have the ability to understand the requirements of the study, provide written informed consent, abide by the study requirements, and agree to return for the required follow-up

Exclusion Criteria:

* failed or incomplete revascularization
* patients with chronic heart failure NYHA IV
* patients with acute coronary syndrome
* patients with severe pulmonary hypertension
* patients who are assigned to conservative PAD treatment (according to the treating physician's decision)
* refusal or inability to give informed consent
* patients who are enrolled into another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PAD patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2009-01 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hehrlein, MD, Study Chair — Department of Cardiology and Angiology, University Hospital of Freiburg, Germany
Locations (1):
- University Hospital of Freiburg, Freiburg im Breisgau, Germany

REFERENCES:
- [Background] Duerschmied D, Olson L, Olschewski M, Rossknecht A, Freund G, Bode C, Hehrlein C. Contrast ultrasound perfusion imaging of lower extremities in peripheral arterial disease: a novel diagnostic method. Eur Heart J. 2006 Feb;27(3):310-5. doi: 10.1093/eurheartj/ehi636. Epub 2005 Nov 24. PMID 16308326